CLINICAL TRIAL: NCT07303829
Title: Laproscopic Managment of Pyogenic Liver Abscess
Brief Title: Laparoscopic Approach to Pyogenic Liver Abscess
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebram Nashat Bastawroos Zakaria, Doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMPLA
Record Dates: First submitted 2025-11-20; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Liver Abscess, Pyogenic
MeSH Terms: conditions — Liver Abscess, Pyogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laproscopic managment (Experimental)
  Interventions: Device: Laproscopic

INTERVENTIONS:
Device: Laproscopic — Laparoscopic management uses minimally invasive trocar access with camera-guided drainage and debridement, allowing precise abscess evacuation, reduced tissue trauma, faster recovery, and lower postoperative pain compared with open surgery or percutaneous drainage used in other studies.

SUMMARY:
Assess the efficacy and safety of laparoscopic management of liver abscess in achieving complete drainage and clinical recovery compared to conventional open or percutaneous methods, and to:

1. To evaluate postoperative complications and recurrence rates.
2. To compare hospital stay, recovery time, and overall morbidity.
3. To determine patient outcomes and cost-effectiveness of laparoscopic intervention.

DETAILED DESCRIPTION:
Liver abscess is a localized collection of pus within the liver parenchyma, most commonly resulting from bacterial or amoebic infection. It remains a serious clinical condition requiring timely diagnosis and effective management to prevent complications such as sepsis or rupture. Traditionally, open surgical drainage was the standard treatment for complicated or multiloculated abscesses and in cases where percutaneous drainage failed. However, advances in minimally invasive surgery have introduced laparoscopic drainage as a safer and more efficient alternative.

Laparoscopic management offers several advantages, including smaller incisions, reduced postoperative pain, shorter hospital stays, and faster recovery compared to open surgery. Moreover, it allows direct visualization of the abscess cavity, facilitates breaking of loculations, debridement of necrotic tissue, and precise placement of drainage catheters. These features enhance the completeness of drainage and reduce recurrence rates.

Recent studies have demonstrated the efficacy of laparoscopic drainage, particularly in large, complex, or multiloculated liver abscesses where percutaneous methods are unsuccessful or contraindicated. A meta-analysis of 17 studies involving 608 patients reported a recurrence rate of only 4.22% with no procedure-related mortality in the laparoscopic group. Consequently, laparoscopic drainage is now considered a step-up approach in the management algorithm of liver abscess, bridging the gap between percutaneous and open surgical techniques, while ensuring optimal clinical outcomes and reduced morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years.
2. Radiologically confirmed liver abscess (US/CT/MRI).
3. Abscess requiring drainage ≥5 cm,
4. Failed or contraindicated percutaneous drainage.
5. Recurrence after percutaneous drainage.

Exclusion Criteria:

1. Adults ≥18 years.
2. Radiologically confirmed liver abscess (US/CT/MRI).
3. Abscess requiring drainage ≥5 cm,
4. Failed or contraindicated percutaneous drainage.
5. Recurrence after percutaneous drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Major complication rate | 30 days
  Procedure-related complications (Clavien-Dindo ≥ III) within 30 days.
Abscess recurrence | 6 months.
  Recurrence at the same or new site

SECONDARY OUTCOMES:
Technical success | 30days
  Successful laparoscopic drainage and drain placement

REFERENCES:
- [Result] Ndong A, Tendeng JN, Diallo AC, Dieye A, Diao ML, Diallo S, Diop S, Diallo MK, Diedhiou M, Fall ML, Ma Nyemb PM, Konate I. Efficacy of laparoscopic surgery in the treatment of hepatic abscess: A systematic review and meta-analysis. Ann Med Surg (Lond). 2022 Jan 31;75:103308. doi: 10.1016/j.amsu.2022.103308. eCollection 2022 Mar. PMID 35198179
- [Result] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Result] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Result] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharm Stat. 2005;4(4):287-291.
- [Result] International Journal of Surgery. Laparoscopic Drainage of Pyogenic Liver Abscess: A Feasible Alternative. https://www.ijsurgery.com/index.php/isj/article/view/9473
- [Result] Bansal V, et al. Systematic Review of Laparoscopic Drainage of Liver Abscess. Cureus. 2022;14(2):e22045. https://pmc.ncbi.nlm.nih.gov/articles/PMC8850317
- [Result] Saravanan R, et al. Comparative Study of Laparoscopic Versus Open Surgical Drainage in Pyogenic Liver Abscess. SAR J Surg. 2024. https://sarpublication.com/media/articles/SARJS_62_10-14.pdf
- [Result] Medscape. Liver Abscess Treatment & Management. https://emedicine.medscape.com/article/188802-treatment